CLINICAL TRIAL: NCT01476124
Title: A Double-Blind, 3-Part Crossover Study to Assess the Pharmacokinetics and Tolerability of Single Doses of Gabapentin Enacarbil and Morphine Administered Alone and in Combination in Healthy Subjects
Brief Title: Drug Drug Interaction Study With Gabapentin Enacarbil and Morphine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115720
Record Dates: First submitted 2011-08-25; First posted 2011-11-22 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2011-11

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen A (Experimental): Morphine placebo + GEn 600 mg
  Interventions: Drug: morphine Placebo; Drug: GEn 600 mg
- Regimen B (Experimental): Morphine Extended release (60 mg) + GEn placebo
  Interventions: Drug: Morphine; Drug: GEn Placebo
- Regimen C (Experimental): Morphine Extended release (60mg) + GEn 600 mg
  Interventions: Drug: GEn 600 mg; Drug: Morphine

INTERVENTIONS:
Drug: morphine Placebo — Morphine Placebo
  Arms: Regimen A
Drug: GEn 600 mg — Gabapentin enacarbil 600 mg
  Other Names: XP13512; GSK1838262
  Arms: Regimen A; Regimen C
Drug: Morphine — morphine extended release 60 mg
  Arms: Regimen B; Regimen C
Drug: GEn Placebo — Gabapentin enacarbil placebo
  Arms: Regimen B

SUMMARY:
This double-blind study will evaluate the pharmacokinetics of a single dose of morphine or gabapentin derived from gabapentin enacarbil (GEn) after administration of morphine and GEn alone and in combination as well as the tolerability of morphine administered with GEn. The dose of GEn will be 600 mg administered with food. Morphine/morphine placebo will be administered 2 hours prior to GEn/GEn placebo in the fasted state. A 60 mg dose of a controlled release formulation of morphine will be given. Blood samples for evaluation of gabapentin, morphine and morphine-6-glucuronide will be collected. The pharmacodynamic effect of co-administering both treatments will be assessed using visual analog scales for somnolence/sedation, dizziness and nausea.

DETAILED DESCRIPTION:
This double-blind study will evaluate the pharmacokinetics of a single dose of morphine or gabapentin derived from gabapentin enacarbil (GEn) after administration of morphine and GEn alone and in combination as well as the tolerability of morphine administered with GEn. The dose of GEn will be 600 mg administered with food. Morphine/morphine placebo will be administered 2 hours prior to GEn/GEn placebo in the fasted state. A 60 mg dose of a controlled release formulation of morphine will be given. Blood samples for evaluation of gabapentin, morphine and morphine-6-glucuronide will be collected. The pharmacodynamic effect of co-administering both treatments will be assessed using visual analog scales for somnolence/sedation, dizziness and nausea.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, clinical laboratory tests, and 12 lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Subject is a male between 18 and 65 years of age inclusive, at the time of signing the informed consent
* Subject has a body weight >55 kg and body mass index (BMI) within the range of 19 to 30 kg/m2 (inclusive)
* Subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form
* Subject has a QTcB <450 ms
* Subject has a creatinine clearance (CrCl) >80 mL/min. The CrCl is estimated using the Cockcroft and Gault equation. Details on CrCl calculations are provided in the Study Procedures Manual (SPM)
* Subject has an aspartate aminotransferase (AST), ALT, and alkaline phosphatase within reference range at the screening visit. Isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35% of the total bilirubin

Exclusion Criteria:

* Subject has positive prestudy drug or alcohol screen results. At minimum, the drug screen will include alcohol, cotinine, amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines
* Subject has positive prestudy (within 3 months of Screening) hepatitis B surface antigen or positive hepatitis C antibody results
* Subject has a positive prestudy human immunodeficiency virus (HIV) antibody result
* Subject has a history of regular alcohol consumption within 6 months of the study defined as: an average intake of >14 drinks/week . One drink is equivalent to (12 g of alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Subject has participated in a clinical trial and has received an investigational product within the following time period before the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Subject has been exposed to more than 4 new chemical entities within 12 months before the first dosing day
* Subject has used prescription or nonprescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study treatment, unless in the opinion of the investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Subject has a history of sensitivity to gabapentin, morphine, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates participation in the study
* Subject's participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period
* Subject is unwilling or unable to follow the procedures outlined in the protocol
* Subject has a screening heart rate <45 or >100 bpm, systolic blood pressure >140 or <100 mm Hg, or diastolic blood pressure >90 or <60 mm Hg in the semi supine position and the value(s) do not return to within reference range upon retest.
* Subject has postural hypotension demonstrated at the screening medical ( defined as a fall in systolic pressure of 30mmHg or more and/or a fall in diastolic pressure of 20mmHg or more after standing for 3 minutes) or a history of clinically significant symptomatic postural hypotension or vaso vagal episodes
* Subject smokes more than 5 cigarettes or equivalent/day. Subjects should continue their smoking/non-smoking habits throughout the study apart from refraining from smoking on study days
* Subject has a history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, GI, endocrine, immunologic, dermatologic, neurologic or psychiatric disease
* Subject has a history of seizures other than febrile seizures as a child
* Subject has received any medications known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration, in the opinion of the Sponsor or investigator
* Subject has a creatine kinase value greater than the ULN that is not explainable by recent strenuous exercise and the value does not return to within reference range upon retest.
* Subject has current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subject is mentally or legally incapacitated
* Subject has a history of respiratory depression, acute or severe bronchial asthma, or hypercarbia
* Subject has or is suspected of having paralytic ileus or chronic constipation
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 7 days
  evaluate the pharmacokinetics of morphine, morphine-6-glucuronide and of gabapentin derived from GEn following administration of single doses of morphine (60 mg) and GEn (600 mg) alone and in combination

SECONDARY OUTCOMES:
Profile of Pharmacokinetics | predose,1,2,3,4,5,6,7,8,9,10,11,12,14,16,18,20,24,26,and 36 hours post dose
  Area under the curve (AUC), Concentration Max (Cmax)
Safety of Patients treated with Gen | Screening to follow-up
  Laboratory safety tests including blood chemistry, urine analysis, ECG testing, and liver enzyme tests

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- [Derived] Chen C, Upward J, Arumugham T, Stier B, Davy M. Gabapentin enacarbil and morphine administered in combination versus alone: a double-blind, randomized, pharmacokinetic, and tolerability comparison. Clin Ther. 2015 Feb 1;37(2):349-57. doi: 10.1016/j.clinthera.2014.10.015. Epub 2014 Nov 20. PMID 25467190